CLINICAL TRIAL: NCT03151928
Title: Diagnostic Accuracy By Providers Study
Acronym: DAP
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Becton Dickinson Life Sciences (Unknown)
Responsible Party: Principal Investigator, Sharon Hillier, Professor, University of Pittsburgh
Other Study IDs: PRO17030332
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Vaginitis
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women presenting with vaginitis symptoms: Women with vaginitis seeking routine care will be approached to have five additional swabs collected during their pelvic exam
  * vaginal swab for qualitative PCR using the BD Max Vaginal Panel on the automated BDMAX System
  * Vaginal smear for evaluation with Gram's stain and Nuget's criteria
  * Vaginal swab for yeast culture
  * Vaginal swab for Trichomonas vaginalis NAAT
  * Vaginal swab for discrepant analysis testing
  Interventions: Diagnostic Test: BDMax Vaginal Panel

INTERVENTIONS:
Diagnostic Test: BDMax Vaginal Panel — The tests will be used to compare results between clinician diagnosis/routine care testing and the above interventions
  Other Names: Gram Stain/Nuget Criteria; yeast culture; Trichomonas vaginalis NAAT

SUMMARY:
The validation study is intended to provide comparative data on the diagnosis of vaginal infections as performed in primary care settings versus the diagnosis provided through standard diagnostic testing performed in a reference laboratory. The clinician and lab diagnoses will be compared to those obtained using the BD MAX Vaginal Panel on the BD MAX System.

DETAILED DESCRIPTION:
The primary goals of this study are to:

1. Compare the level of agreement of clinician diagnosed bacterial vaginosis (BV) to vaginal swab samples evaluated for BV using Nugent's criteria and the BD MAX Vaginal Panel
2. Compare the level of agreement of clinician diagnosed trichomonas vaginalis (TV) to the laboratory diagnosis of TV identified by quantitative PCR using the GeneXpert system by Cepheid and the BD MAX Vaginal Panel.
3. Compare the level of agreement of clinician diagnosed yeast vaginitis to laboratory diagnosis of yeast identified with culture and the BD MAX Vaginal Panel.

The secondary goals of this study include:

1. Being able to describe the patterns of testing among clinicians in community practices providing routine care for women presenting with symptoms of vaginitis.
2. Describe the treatments prescribed for women presenting with vaginitis and how these prescribed treatments are distributed in women with laboratory-confirmed diagnoses.

ELIGIBILITY:
Inclusion Criteria:

1. Female, Age 18-40
2. Presenting with symptoms of vaginitis; vaginal discharge, vaginal odor, vulvar or vaginal itch, vulvar or vaginal discomfort (i.e. irritation, burning pain or vulvar edema).
3. Able and willing to provide verbal consent.
4. Willingness to undergo all study-related assessments and procedures, including the collection of multiple vaginal swabs, answer questions related to demographic and health information and follow all other study-related procedures.

Exclusion:

Women who meet any of the following criteria by participant report will be excluded from the study:

1.) Any condition that, in the opinion of the Investigator, would preclude provision of consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Study Population: Women presenting to primary care offices with symptoms of vaginitis
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
BV Result Agreement | enrollment
  Comparison of the level of agreement of clinician diagnosed BV to vaginal swab samples evaluated for BV using Nugent's criteria and the BD MAX Vaginal Panel
Trichomonas (TV) Result Agreement | enrollment
  Comparison of the level of agreement of clinician diagnosed TV to the laboratory diagnosis of TV identified by quantitative PCR using the GeneXpert system by Cepheid and the BD MAX Vaginal Panel
Yeast Result Agreement | enrollment
  Comparison of the level of agreement of clinician diagnosed yeast vaginitis to laboratory diagnosis of yeast identified with culture and the BD MAX Vaginal Panel

SECONDARY OUTCOMES:
Patterns of clinician testing | enrollment
  Description of the patterns of testing among clinicians in the community practice providing care for women presenting with symptoms of vaginitis
Prescribed Treatments | enrollment
  Description of the treatments prescribed for women presenting with vaginitis and how these prescribed treatments are distributed in women with laboratory confirmed diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Hillier, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC/associated community clinics, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hillier SL, Austin M, Macio I, Meyn LA, Badway D, Beigi R. Diagnosis and Treatment of Vaginal Discharge Syndromes in Community Practice Settings. Clin Infect Dis. 2021 May 4;72(9):1538-1543. doi: 10.1093/cid/ciaa260. PMID 32350529